CLINICAL TRIAL: NCT05111444
Title: Camrelizumab Plus Pyrotinib Plus Chemotherapy in Human Epidermal Growth Factor Receptor 2 Positive (HER2+) Advanced Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-SH-GC-II-010
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Gastric Neoplasms; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; pyrotinib; Capecitabine; Oxaliplatin; Paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Pyrotinib + Chemotherapy (Other): Camrelizumab (200 mg) will be administered intravenously [IV] on day 1 of each 3-week cycle. Pyrotinib (320 mg) will be administered orally once daily [QD] on every 21 days. Chemotherapy will either be XELOX, SOX or TS.
  Interventions: Drug: Camrelizumab; Drug: Pyrotinib; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Paclitaxel; Drug: S-1

INTERVENTIONS:
Drug: Camrelizumab — 200 mg on Day 1 of each 3-week cycle as an IV infusion
Drug: Pyrotinib — 320mg as continuous oral once daily on every 21 days
Drug: Capecitabine — 1000 mg/m^2 as oral capsules BID on Days 1-14 of each 3-week cycle, administered as part of XELOX chemotherapy regimen
Drug: Oxaliplatin — 130 mg/m^2 on Day 1 of each 3-week cycle over 2 hours as an IV infusion, administered as part of XELOX chemotherapy regimen and as part of SOX chemotherapy regimen
Drug: Paclitaxel — 80 mg/m^2 on Day 1 and Day 8 of each 3-week cycle as an IV infusion, administered as part of FP chemotherapy regimen
Drug: S-1 — Combination product of tegafur, CDHP, and Oxo. Oral capsules BID on Days 1-14 of each 3-week cycle based on body surface area (BSA): <1.25 m^2 BSA =40 mg, 1.25 to <1.5 m^2 BSA=50 mg, ≥1.5 m^2 BSA=60 mg. Administered as part of SOX and TS chemotherapy regimen

SUMMARY:
This study is designed to evaluate the efficacy and safety of Camrelizumab plus pyrotinib in combination with chemotherapy in patients with HER2-positive gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Histologically or cytologically confirmed diagnosis of locally advanced unresectable or metastatic HER2 positive gastric or GEJ adenocarcinoma.
3. Patients have not received systemic treatment in the past but had disease progression more than 6 months after receiving neoadjuvant therapy or the last of adjuvant therapy could be enrolled or failure of first-line therapy or completion of (new) adjuvant therapy to disease recurrence less than 6 months.
4. HER2-positive defined as either immunohistochemistry (IHC) 3+ or IHC 2+ in combination with fluorescent in-situ hybridization (FISH+ is defined as HER2:CEP17 ratio≥2.0), as assessed by central review on primary or metastatic tumor.
5. ECOG performance status 0-1.
6. At least one measurable lesion exists as defined by RECIST 1.1 .
7. Life expectancy of more than 12 weeks.

Exclusion Criteria:

1. Hypersensitivity to Camrelizumab, pyrotinib and study chemotherapy agents and/or to any components.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40, Cluster of Differentiation 137 [CD137]).
3. Has an active autoimmune disease that has required systemic treatment in past 2 years.
4. Has a known history of Human Immunodeficiency Virus (HIV) or active hepatitis B and C virus infection.
5. Has had major surgery within 28 days prior to randomization, or anticipation of the need for major surgery during the course of study treatment.
6. Subjects who can not interrupt the using of the drugs that may cause QT prolongation during study.
7. Evidence or history of coagulation disorders such as a grade ≥ 3 (CTC-AE) bleeding event.
8. Known history of psychotropic substance abuse or drug use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | [ Time Frame: Up to approximately 2 years ]
  Objective response rate assessed at 18 weeks after enrollment，that is about 6 cycles of treatment

SECONDARY OUTCOMES:
Progression Free Survival (PFS) per RECIST 1.1 assessed by BICR | [ Time Frame: Up to approximately 2 years ]
  The time from the beginning of treatment to the progression or death of the patient
Overall Survival (OS) | [ Time Frame: Up to approximately 2 years ]
  The time from the beginning of treatment to the death of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- 270 Dongan Road, Fudan University Shanghai Cancer Center, Shanghai, China